CLINICAL TRIAL: NCT03559556
Title: Validation Study of Treating Arteriovenous Malformation With Stereotactic Radiosurgery Using CT Angiography for Treatment Planning
Brief Title: Treating Arteriovenous Malformation With Stereotactic Radiosurgery Using CT Angiography for Treatment Planning
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU 042018-100
Record Dates: First submitted 2018-05-18; First posted 2018-06-18 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Arteriovenous Malformations
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Intervention Model Description: The study proposes to evaluate whether a target volume based on CT angiography can serve as a reliable substitute for a target based on interventional cerebral arteriography. Patients on this protocol will still get treated based on target generated by interventional cerebral arteriography but also receive CT angiography. If the target volume based on CT angiography are adequate compared to their invasive counterpart, future investigators may selectively omit performing interventional cerebral arteriography in the treatment planning for SRS of AVM. Use of CT angiography may lead to reduction in the risk from the procedure and cost, improve the efficiency of the treatment process ideally without compromising the success of the procedure, with greater patient comfort and satisfaction.
Masking Description: Neurosurgeon who contoured AVM nidus using interventional cerebral arteriography.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with AVM requiring radiotherapy (Experimental): Patients on this protocol will still get treated based on target generated by interventional cerebral arteriography but also receive CT angiography.
  Interventions: Other: CT angiography

INTERVENTIONS:
Other: CT angiography — CT angiography uses a CT scanner to produce detailed images of both blood vessels and tissues in various parts of the body. An iodine-rich contrast material (dye) is usually injected through a small catheter placed in a vein of the arm.

SUMMARY:
Evaluate whether a treatment plan based on CT angiography can accurately and precisely identify the target nidus as compared to standard cerebral arteriography fused to MRI.

DETAILED DESCRIPTION:
Stereotactic Radiosurgery is a preferable treatment option for patients with Arteriovenous malformation (AVM) that are not surgically accessible or in patients with comorbidities that make them poor surgical candidates At University of Texas Southwestern Medical Center (UTSW), investigator routinely perform interventional cerebral arteriography on the day of the SRS procedure for improved target delineation. Even though the addition of angiography is time consuming and requires multi-modality team care, this approach has allowed UTSW to treat the smallest possible target, yet achieve excellent obliteration rates of AVM with very low toxicity from the procedure. At UTSW the investigator also use CT angiogram at the treatment team's discretion to further enhance the accurate delineation of the final treatment target volume. However, it had not been routinely done due to uncertain benefit in treatment planning and a concern for renal burden from additional intravenous (IV) contrast usage.

This prospective enrollment and conduct open-label, retrospective analysis study is to evaluate whether a target volume based on CT angiography can serve as a reliable substitute for a target based on interventional cerebral arteriography. Patients on this protocol will still get treated based on target generated by interventional cerebral arteriography but also receive CT angiography. If the target volume based on CT angiography are adequate compared to their invasive counterpart, future investigators may selectively omit performing interventional cerebral arteriography in the treatment planning for SRS of AVM. Use of CT angiography may lead to reduction in the risk from the procedure and cost, improve the efficiency of the treatment process ideally without compromising the success of the procedure, with greater patient comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Documented AVM with draining vein(s).
2. Adequate renal function (serum Creatinine < 1.5 mg/dl within 30 days of SRS) to undergo contrast CT and interventional cerebral arteriography on the same day, as determined by treating physicians.
3. AVM must be physically separated from the optic pathway, brainstem or spinal cord.
4. The maximum diameter of AVM nidus must be less than 3.5 cm and/or less than 12 cc.
5. Age ≥ 10 years.
6. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

   6.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
7. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Patients without a documented AVM.
2. Patients with a contraindication to CT or MRI such as contrast allergy, kidney failure or implanted metal devices or foreign bodies or severe claustrophobia.
3. Use of Nephrotoxic drugs, such as gentamycin, high-dose nonsteroidal anti-inflammatory drugs, or certain chemotherapeutic drugs within 10 days of the procedure.
4. Psychiatric illness/social situations that would limit compliance with study requirements.
5. Patients must not be pregnant at the time of SRS treatment.

Ages: 10 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient With AVM Requiring Radiotherapy: Patients who received planning CT angiogram in addition to standard of care
  CT angiography: CT angiography uses a CT scanner to produce detailed images of both blood vessels and tissues in various parts of the body. An iodine-rich contrast material (dye) is usually injected through a small catheter placed in a vein of the arm.
Period: Overall Study
Arm/Group | Patient With AVM Requiring Radiotherapy
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled to study
Arm/Group | Patient With AVM Requiring Radiotherapy
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Target Volume Difference Between Standard of Care vs. CT Angiogram and MRI Alone
Description: The primary endpoint of this study is to compare the volumes of targets generated from interventional cerebral arteriography (reference) to targets generated from CT angiogram and MRI alone, to assess whether noninvasive imaging approaches are noninferior to the UTSW standard
Time Frame: Same day measurements
Population: Median volume between standard of care target volumes (mL) vs. CT Angiogram in addition to standard of care. Standard of care is considered reference volume
Measure: Median (Standard Deviation); unit: mL
Groups:
- CT Angiogram in Addition to Standard of Care: Patients who received planning CT angiogram in addition to standard of care
- Standard of Care: Standard of Care MRI and IR angiogram
Arm/Group | CT Angiogram in Addition to Standard of Care | Standard of Care
Number analyzed (Participants) | 13 | 13
mL | 1.1 (2.5) | 1.3 (2.4)

2. Secondary Outcome: CT Angiogram Additional Time
Description: Additional time required for CT angiogram after standard of care imaging
Time Frame: Same day
Population: Time required for CT angiogram
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Additional Time Required for CT Angiogram: Patients who received planning CT angiogram in addition to standard of care
Arm/Group | Additional Time Required for CT Angiogram
Number analyzed (Participants) | 13
Minutes | 8 (4.3)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Patient With AVM Requiring Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient With AVM Requiring Radiotherapy (N=13)
urine discoloration (Renal and urinary disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03559556/Prot_SAP_000.pdf